CLINICAL TRIAL: NCT07364994
Title: Effectiveness of a Team Based Learning Intervention on Evidence-Based Practice Competence Among Nursing Students: A Quasi-Experimental Study
Brief Title: Effectiveness of a Team-Based Learning Intervention on Evidence-Based Practice Competence Among Nursing Students.
Acronym: TBL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Paola Ferri, Associate Professor MEDS-24/C General, Clinical, Pediatric, Obstetric-Gynecological, and Neonatal Nursing Sciences Chair of the Nursing Degree Program in Modena, University of Modena and Reggio Emilia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FINE-EU-2026
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Nursing Education in Evidence-Based Practice; Active Learning Methods and Life-skills Education; Evidence Based Nursing; Evidence Based Programs in Schools; Nursing Education; Evidence Based Practice; Education Advancement; Education, Competency-Based; Education, Nursing Students
Keywords: Evidence-Based Practice; Nursing Education; Curriculum; Learning; Problem-Based Learning; Team-Based Learning; Flipped Classroom; Critical Thinking; Competency-Based Education; Active Learning; Self Efficacy
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, single-cohort, pre-test/post-test design. All participants received the composite educational intervention (Flipped Classroom + Team-Based Learning). There was no concurrent control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBP Educational Intervention Arm (Experimental): Single cohort of second-year nursing students receiving the composite educational intervention.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — A structured, credit-bearing educational module on Evidence-Based Practice (EBP) integrated into a 64-hour course. The experimental intervention specifically targets the 'Core EBP' component (12 contact hours), delivered exclusively via Team-Based Learning (TBL) by an experienced academic facilitator with expertise in nursing research and EBP education.
  The intervention follows the structured TBL cycle across three in-person sessions of 4 hours each:
  * Individual Preparation: Prior to sessions, students engage in self-directed study of preparatory scientific articles and lecture notes.
  * Readiness Assurance Process: Each session begins with an Individual Readiness Assurance Test (iRAT) followed by a Team Readiness Assurance Test (tRAT) with immediate feedback.
  * Appeals and Application: Following an appeals process, the majority of class time is dedicated to application-focused exercises where small, permanent teams solve complex clinical scenariosto support clinical decision-making.
  Other Names: Composite Flipped Classroom and Team-Based Learning (FC-TBL) Programme for EBP

SUMMARY:
The goal of this interventional study is to evaluate the effectiveness of a composite active learning strategy, integrating the Flipped Classroom model and Team-Based Learning (TBL), for improving Evidence-Based Practice (EBP) competence in second-year undergraduate nursing students.

The main questions it aims to answer are:

* Does the educational intervention significantly improve students' self-reported knowledge of EBP concepts?
* Does the educational intervention significantly improve students' self-reported skills in EBP processes (e.g., critical appraisal)?
* Does the educational intervention significantly improve students' attitudes towards EBP?

Participants, who were all second-year nursing students enrolled in a specific academic year, took part in a mandatory 64-hour EBP educational module. Their main tasks were:

* To complete a validated self-assessment questionnaire (the Evidence-Based Practice Competence Questionnaire, EBP-COQ) at baseline (March 2024) and immediately following the intervention (April 2024).
* To engage in the "Core EBP" module of the course (12 hours), which was delivered using a Team-Based Learning (TBL) strategy. This module comprised:
* Asynchronous individual preparatory study (Flipped Classroom phase) of provided scientific articles and lecture notes, conducted 1-2 weeks prior to each session.
* Participation in three in-person, 4-hour interactive sessions (12 contact hours total), following the structured TBL cycle of Readiness Assurance (iRAT and tRAT) and Team Application exercises.

DETAILED DESCRIPTION:
1. Background and Rationale

   Evidence-Based Practice (EBP) is a fundamental competency for healthcare professionals, integral to delivering high-quality, safe, and effective patient care. International nursing organisations and educational frameworks consistently mandate the integration of EBP competencies into undergraduate curricula. However, significant variability persists in how EBP is taught, with traditional, lecture-based methods often proving insufficient for developing the complex skills required for its application in clinical practice.

   Contemporary educational research advocates for active, student-centred learning strategies to effectively teach EBP. The Flipped Classroom (FC) model and Team-Based Learning (TBL) are two such pedagogies. FC facilitates preparatory acquisition of foundational knowledge, thereby liberating in-class time for higher-order learning activities. TBL provides a structured framework for applying knowledge through collaborative problem-solving, critical discussion, and peer feedback, which are essential for mastering EBP steps like critical appraisal and clinical integration.

   While the individual effectiveness of FC and TBL has been explored, there is a paucity of research evaluating a structured, composite intervention that sequentially combines these methodologies specifically to enhance EBP competence in nursing students within a European context. This study aims to address this gap.
2. Study Design and Setting

   This is a quasi-experimental, single-centre study employing a pre-test/post-test design without a control group. The study was conducted within the Bachelor of Nursing degree programme at the University of Modena and Reggio Emilia (Modena site), Italy.

   The target population was the entire cohort of second-year nursing students enrolled in the academic year 2023-2024. This stage was selected as students begin to synthesise theoretical knowledge with clinical practice, representing a pivotal point for EBP skill development.
3. Participant Recruitment and Ethical Considerations

   All eligible students were invited to participate. The study protocol, including participant information sheets and consent forms, was reviewed and approved by the Institutional Ethical Committee for Research (CEAR) of the University of Modena and Reggio Emilia prior to commencement. Participation was entirely voluntary, and written informed consent was obtained from all participants. Refusal to participate did not affect academic standing or access to the educational module.

   To ensure confidentiality and data protection, a strict anonymisation procedure was implemented. Participants created a unique personal code to link their pre- and post-intervention questionnaires, ensuring no directly identifiable data was stored with the research data.
4. Detailed Description of the Educational Intervention

   The intervention was a dedicated, credit-bearing EBP module integrated into a broader 64-hour "Evidence-Based Nursing" course within the second-year curriculum. The experimental intervention specifically targeted the Core EBP module (12 contact hours), delivered exclusively using a Team-Based Learning (TBL) strategy.

   Teaching Team: The module was delivered by a single experienced academic with an established track record in EBP pedagogical research.

   Pedagogical Model: Team-Based Learning (TBL).

   Pre-Session (FC Phase): One to two weeks prior to each in-person session, students engaged with preparatory materials (e.g., selected scientific articles and specific lecture notes) hosted on the university's Moodle platform.

   In-Session (TBL Phase): The intervention consisted of three 4-hour sessions (12 contact hours total) conducted over a five-week period. Sessions were structured according to TBL principles:
   * Readiness Assurance Process: Each session began with a 10-item multiple-choice Individual Readiness Assurance Test (iRAT), followed by the same test taken in permanent, instructor-formed teams (tRAT). Immediate feedback was provided via the Immediate Feedback Assessment Technique (IF-AT).
   * Appeals Process: Teams could submit written justifications to challenge test questions, requiring consultation of the preparatory materials.
   * Application-Focused Exercises: The majority of each session (2.5 to 3 hours) was dedicated to solving complex clinical cases. These exercises followed the "4 S" framework (Significant Problem, Same Problem, Specific Choice, and Simultaneous Report) to practice formulating PICO questions, bibliographic searching, appraising research articles, and integrating evidence into clinical decision-making.
5. Outcome Measurement and Data Collection

   The primary outcome was the change in self-reported EBP competence, measured using the validated Italian version of the Evidence-Based Practice Competence Questionnaire (EBP-COQ). The instrument assesses three domains: Attitudes (13 items), Skills (6 items), and Knowledge (6 items), using a 5-point Likert scale.

   Data collection occurred at two time points:
   * Pre-test (T0): Administration of the EBP-COQ during the recruitment and baseline phase on 4th March 2024.
   * Post-test (T1): Administration of the EBP-COQ immediately following the final session on 22nd April 2024.
6. Statistical Methods

Data analysis will be perform using statistical software (SPSS, version 27.0). Descriptive statistics will summarise participant characteristics. The primary analysis will involve paired-sample t-tests to compare mean scores for the total EBP-COQ and its three subscale scores (Attitudes, Skills, Knowledge) between T0 and T1. The threshold for statistical significance will beset at p < 0.05. To estimate the magnitude of change, Cohen's d effect sizes will be calculate for significant comparisons. Sensitivity analysis will be performed using Wilcoxon signed-rank test. The relationship between individual preparation (iRAT) and team gain (tRAT-iRAT) will be assessed via Spearman's correlation, to evaluate the collaborative learning impact. Data will be handle using a complete-case analysis strategy (listwise deletion).

ELIGIBILITY:
Inclusion Criteria:

* Being a Nursing Student
* Enrolled as a second-year student in the Bachelor of Nursing degree at the study site (University of Modena and Reggio Emilia, Modena campus) for the 2023-2024 academic year.
* Attended the first lecture of the course where the study was presented (or were otherwise fully informed about it).
* Provided written informed consent to participate in the research.

Exclusion Criteria:

* Not formally enrolled in the second year of the Nursing programme at the study site for the 2023-2024 academic year.
* Had already obtained recognition/validation of the academic credit for the specific Evidence-Based Practice (EBP) course unit before the study began.
* Were absent for the entire duration of the EBP educational module.
* Declined to give informed consent to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Overall Evidence-Based Practice Competence Score | Baseline (T0, pre-intervention) and Post-intervention (T1, at the completion of the educational module, approximately 2 months after baseline).
  The overall competence in Evidence-Based Practice (EBP) is measured using the validated Italian version of the Evidence-Based Practice Competence Questionnaire (EBP-COQ). This is a self-reported questionnaire consisting of 25 items rated on a 5-point Likert scale (1=Strongly Disagree to 5=Strongly Agree). The Overall Score is calculated as the sum of the scores from all 25 items. Total Score Range: 25 - 125. A higher total score indicates a higher self-perceived competence in EBP. The change in the Overall Score from baseline (T0) to post-intervention (T1) is the primary outcome.

SECONDARY OUTCOMES:
EBP Attitude Domain Score | Baseline (T0, pre-intervention) and Post-intervention (T1, at the completion of the educational module, approximately 2 months after baseline).
  Score for the Attitude domain of the Evidence-Based Practice Competence Questionnaire (EBP-COQ). This domain comprises 13 items assessing beliefs, perceptions, and values regarding the usefulness and application of EBP in nursing (e.g., "EBP helps in making clinical decisions"). The score is the sum of these 13 items (score range 13 - 65). A higher score indicates a more positive attitude towards EBP.
EBP Skills/Competence Domain Score | Baseline (T0, pre-intervention) and Post-intervention (T1, at the completion of the educational module, approximately 2 months after baseline).
  Score for the Skills/Competence domain of the Evidence-Based Practice Competence Questionnaire (EBP-COQ). This domain comprises 6 items assessing the self-perceived ability to to perform key EBP steps like critically evaluating and applying research evidence (e.g., "I feel able to critically assess the quality of a scientific article"). The score is the sum of these 6 items (score range 6 - 30). A higher score indicates greater perceived skill in executing EBP processes.
EBP Knowledge Domain Score | Baseline (T0, pre-intervention) and Post-intervention (T1, at the completion of the educational module, approximately 2 months after baseline).
  Score for the Knowledge domain of the Evidence-Based Practice Competence Questionnaire (EBP-COQ). This domain comprises 6 items assessing knowledge of key EBP principles and understanding of research methodologies (e.g., knowledge of PICO framework, levels of evidence, main study designs). The score is the sum of these 6 items (score range 6 - 30). A higher score indicates greater self-assessed knowledge of EBP concepts.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Ferri, MSc, Principal Investigator — University of Modena and Reggio Emilia; Teresa Peduto, MSc, Study Chair — Azienda Ospedaliero-Universitaria di Modena; Angela Contri, PhD, Study Chair — University of Modena and Reggio Emilia
Locations (1):
- University of Modena and Reggio Emilia, Modena, Missouri, Italy

IPD SHARING:
Plan to Share IPD: No
The Individual Participant Data (IPD) collected for this study contains detailed and sensitive personal information. To ensure the confidentiality and privacy of our participants in compliance with stringent EU and Italian data protection regulations (GDPR), the data will not be made publicly available. The data will be kept securely within the institutional responsibility of the University of Modena and Reggio Emilia for the purposes outlined in this protocol.

REFERENCES:
- [Background] Ramos-Morcillo AJ, Fernandez-Salazar S, Leal-Costa C, Ruzafa-Martinez M. Evidence-based practice nurses' competency: Spanish national survey and establishment of a scale of the EBP-COQ-Prof(c). J Nurs Manag. 2021 May;29(4):794-804. doi: 10.1111/jonm.13220. Epub 2020 Dec 20. PMID 33259110
- [Background] Tlili MA, Aouicha W, Tarchoune S, Sahli J, Ben Dhiab M, Chelbi S, Mtiraoui A, Ajmi T, Ben Rejeb M, Mallouli M. Predictors of evidence-based practice competency among Tunisian nursing students. BMC Med Educ. 2022 Jun 2;22(1):421. doi: 10.1186/s12909-022-03487-4. PMID 35655300
- [Background] Straus SE, Glasziou P, Richardson WS, Haynes RB. Evidence-based Medicine E-Book: How to Practice and Teach EBM; Elsevier Health Sciences: Amsterdam, The Netherlands, 2018.
- [Background] Stichler JF, Fields W, Kim SC, Brown CE. Faculty knowledge, attitudes, and perceived barriers to teaching evidence-based nursing. J Prof Nurs. 2011 Mar-Apr;27(2):92-100. doi: 10.1016/j.profnurs.2010.09.012. PMID 21420041
- [Background] Skela-Savic B, Gotlib J, Panczyk M, Patelarou AE, Bole U, Ramos-Morcillo AJ, Finotto S, Mecugni D, Jarosova D, Patelarou E, Dolezel J, Ruzafa-Martinez M. Teaching evidence-based practice (EBP) in nursing curricula in six European countries-A descriptive study. Nurse Educ Today. 2020 Nov;94:104561. doi: 10.1016/j.nedt.2020.104561. Epub 2020 Aug 27. PMID 32905986
- [Background] Sackett DL, Rosenberg WM, Gray JA, Haynes RB, Richardson WS. Evidence based medicine: what it is and what it isn't. BMJ. 1996 Jan 13;312(7023):71-2. doi: 10.1136/bmj.312.7023.71. No abstract available. PMID 8555924
- [Background] Ruzafa-Martinez M, Fernandez-Salazar S, Leal-Costa C, Ramos-Morcillo AJ. Questionnaire to Evaluate the Competency in Evidence-Based Practice of Registered Nurses (EBP-COQ Prof(c)): Development and Psychometric Validation. Worldviews Evid Based Nurs. 2020 Oct;17(5):366-375. doi: 10.1111/wvn.12464. Epub 2020 Oct 22. PMID 33089629
- [Background] Ruzafa-Martinez M, Molina-Rodriguez A, Perez-Munoz V, Leal-Costa C, Ramos-Morcillo AJ. Effectiveness of the flipped classroom methodology on the learning of evidence-based practice of nursing students: Quasi-experimental design. Nurse Educ Today. 2023 Sep;128:105878. doi: 10.1016/j.nedt.2023.105878. Epub 2023 Jun 18. PMID 37352765
- [Background] Ruzafa-Martinez M, Lopez-Iborra L, Moreno-Casbas T, Madrigal-Torres M. Development and validation of the competence in evidence based practice questionnaire (EBP-COQ) among nursing students. BMC Med Educ. 2013 Feb 7;13:19. doi: 10.1186/1472-6920-13-19. PMID 23391040
- [Background] Patelarou AE, Mechili EA, Ruzafa-Martinez M, Dolezel J, Gotlib J, Skela-Savic B, Ramos-Morcillo AJ, Finotto S, Jarosova D, Smodis M, Mecugni D, Panczyk M, Patelarou E. Educational Interventions for Teaching Evidence-Based Practice to Undergraduate Nursing Students: A Scoping Review. Int J Environ Res Public Health. 2020 Aug 31;17(17):6351. doi: 10.3390/ijerph17176351. PMID 32878256
- [Background] Parmelee D, Michaelsen LK, Cook S, Hudes PD. Team-based learning: a practical guide: AMEE guide no. 65. Med Teach. 2012;34(5):e275-87. doi: 10.3109/0142159X.2012.651179. Epub 2012 Apr 4. PMID 22471941
- [Background] Pendoni, R., Motta, P. C., Bozzetti, M., & Marcomini, I. (2024). Effectiveness of EBPEPU (evidence-based practice educational program in undergraduate nursing education): a before-after study. Teaching and Learning in Nursing, 19(3), 225-228. https://doi.org/10.1016/j.teln.2024.02.017
- [Background] Palese A, Gonella S, Brugnolli A, Mansutti I, Saiani L, Terzoni S, Destrebecq A, Zannini L, Grassetti L, Dimonte V; SVIAT TEAM. Nursing students' interprofessional educational experiences in the clinical context: findings from an Italian cross-sectional study. BMJ Open. 2019 Mar 20;9(3):e025575. doi: 10.1136/bmjopen-2018-025575. PMID 30898820
- [Background] Mariano C. NURSING EMERGING. ANA Nursing: Scope and Standards of Practice, (2015) 3rd Edition. Beginnings. 2016 Apr;36(2):5, 32-4. PMID 27305802
- [Background] Malik G, McKenna L, Griffiths D. Endeavoring to Contextualize Curricula Within an EBP Framework: A Grounded Theory Study. West J Nurs Res. 2018 Dec;40(12):1765-1784. doi: 10.1177/0193945917753589. Epub 2018 Jan 22. PMID 29357759
- [Background] Leiviska E, Pezaro S, Kneafsey R, Morini L, DeWinter A. Teaching and interconnecting research and evidence-based practice in midwifery and nursing education: A mixed methods systematic review. Nurse Educ Today. 2025 Jul;150:106701. doi: 10.1016/j.nedt.2025.106701. Epub 2025 Mar 17. PMID 40121700
- [Background] Lehane E, Leahy-Warren P, O'Riordan C, Savage E, Drennan J, O'Tuathaigh C, O'Connor M, Corrigan M, Burke F, Hayes M, Lynch H, Sahm L, Heffernan E, O'Keeffe E, Blake C, Horgan F, Hegarty J. Evidence-based practice education for healthcare professions: an expert view. BMJ Evid Based Med. 2019 Jun;24(3):103-108. doi: 10.1136/bmjebm-2018-111019. Epub 2018 Nov 15. PMID 30442711
- [Background] Lam CK, Schubert C. Evidence-Based Practice Competence in Nursing Students: An Exploratory Study With Important Implications for Educators. Worldviews Evid Based Nurs. 2019 Apr;16(2):161-168. doi: 10.1111/wvn.12357. PMID 30977591
- [Background] Labrague LJ, McEnroe-Pettite D, Tsaras K, D'Souza MS, Fronda DC, Mirafuentes EC, Yahyei AA, Graham MM. Predictors of evidence-based practice knowledge, skills, and attitudes among nursing students. Nurs Forum. 2019 Apr;54(2):238-245. doi: 10.1111/nuf.12323. Epub 2018 Dec 24. PMID 30582630
- [Background] Kyriakoulis K, Patelarou A, Laliotis A, Wan AC, Matalliotakis M, Tsiou C, Patelarou E. Educational strategies for teaching evidence-based practice to undergraduate health students: systematic review. J Educ Eval Health Prof. 2016 Sep 22;13:34. doi: 10.3352/jeehp.2016.13.34. eCollection 2016. PMID 27649902
- [Background] Kim JS, Gu MO, Chang H. Effects of an evidence-based practice education program using multifaceted interventions: a quasi-experimental study with undergraduate nursing students. BMC Med Educ. 2019 Mar 4;19(1):71. doi: 10.1186/s12909-019-1501-6. PMID 30832639
- [Background] Institute of Medicine (US) Committee on the Robert Wood Johnson Foundation Initiative on the Future of Nursing, at the Institute of Medicine. The Future of Nursing: Leading Change, Advancing Health. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK209880/ PMID 24983041
- [Background] Fiset VJ, Graham ID, Davies BL. Evidence-Based Practice in Clinical Nursing Education: A Scoping Review. J Nurs Educ. 2017 Sep 1;56(9):534-541. doi: 10.3928/01484834-20170817-04. PMID 28876439
- [Background] Finotto S, Garofalo E. [Italian Validation of Evidence Based Practice Evaluation Competence Questionnaire (EBP-COQ)]. Prof Inferm. 2020 Apr-Jun;73(2):98-105. doi: 10.7429/pi.2020.732098. Italian. PMID 33010125
- [Background] Dawes M, Summerskill W, Glasziou P, Cartabellotta A, Martin J, Hopayian K, Porzsolt F, Burls A, Osborne J; Second International Conference of Evidence-Based Health Care Teachers and Developers. Sicily statement on evidence-based practice. BMC Med Educ. 2005 Jan 5;5(1):1. doi: 10.1186/1472-6920-5-1. PMID 15634359
- [Background] Alqahtani N, Oh KM, Kitsantas P, Rodan M. Nurses' evidence-based practice knowledge, attitudes and implementation: A cross-sectional study. J Clin Nurs. 2020 Jan;29(1-2):274-283. doi: 10.1111/jocn.15097. Epub 2019 Nov 26. PMID 31714647
- [Background] Alizadeh M, Masoomi R, Mafinejad MK, Parmelee D, Khalaf RJ, Norouzi A. Team-based learning in health professions education: an umbrella review. BMC Med Educ. 2024 Oct 11;24(1):1131. doi: 10.1186/s12909-024-06147-x. PMID 39394140
- [Background] Alberti S, Motta P, Ferri P, Bonetti L. The effectiveness of team-based learning in nursing education: A systematic review. Nurse Educ Today. 2021 Feb;97:104721. doi: 10.1016/j.nedt.2020.104721. Epub 2020 Dec 11. PMID 33385942
- [Background] Albarqouni L, Hoffmann T, Straus S, Olsen NR, Young T, Ilic D, Shaneyfelt T, Haynes RB, Guyatt G, Glasziou P. Core Competencies in Evidence-Based Practice for Health Professionals: Consensus Statement Based on a Systematic Review and Delphi Survey. JAMA Netw Open. 2018 Jun 1;1(2):e180281. doi: 10.1001/jamanetworkopen.2018.0281. PMID 30646073